CLINICAL TRIAL: NCT00341497
Title: Biomarkers for Oral Cancer
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999998040; OH98-D-N040
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Lichen Planus; Oral Leukoplakia; Mouth Neoplasms
Keywords: Leukoplakia; Oral Mucosa; Biomarkers; Natural History
MeSH Terms: conditions — Lichen Planus; Leukoplakia, Oral; Mouth Neoplasms; Leukoplakia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort: Persons seen at dental clinics at 6 Veterans Affairs Medical Centers who had clinically visibleoral lesions

SUMMARY:
The purpose is to determine the extent of genetic damage in oral mucosal lesions ascertained in the study, whether specific genotypes are associated with genetic damage observed in the oral mucosal lesions, whether the extent of genetic damage changes over time, and what factors (e.g. smoking) contribute to those changes. Genetic damage indicators will include among others DNA adduct formation, particularly related to tobacco smoke carcinogens such as polycyclic aromatic hydocarbons. The genotypes of interest will be focused on these affecting carcinogen metabolism, (e.g., (CYP family), but may also include those related to growth factors, cell cycle control, and DNA repair. Microsatellite instability is another key indicator of damage that we plan to examine. This study was undertaken due to the paucity of data on the types of oral lesions seen in general dental practice and the limited knowledge of the natural history of these lesions.

Persons were enrolled who had red and/or white oral lesions identified at 6 Dental Clinics at VA Medical Centers. The VA Centers involved were: Washington, DC; Atlanta, GA; Durham, NC; San Francisco, CA; Danville, IL; and San Antonio, TX.

When a dentist found a red or white lesions in the course of routine outpatient examinations and care, obvious causes such as denture frictional lesions could be ruled out, and the normal standard of care for the lesion was biopsy, the patient was considered for enrollment into the study. The study was described to the patient, the consent for was signed, the patient received an intraoral examination to identify and characterize the oral lesions, the lesions were photographed, an oral epithelial cell sample was taken from the site and from the rest of the oral mucosa, and the patient was interviewed using a standard questionnaire that requested information about sociodemograhic, medical, and lifestyle factors, particularly tobacco and alcohol use all as part of the study protocol, and the patient received a biopsy as part of normal care. The biopsy report was obtained as was a small piece of the biopsy material that was not needed for patient diagnostic purposes. The subjects returned every 4-6 months for reassessment of the lesion or to determine that the lesion had not returned. The patients completed a questionnaire at each of these visits so that lifestyle factors such as tobacco and alcohol use could be reassessed. Also oral epithelial cell scrapings were obtained at each of these visits.

This study is particularly valuable because longitudinal data was collected and because the data were collected over time using standard procedures.

DETAILED DESCRIPTION:
This longitudinal research project is part of a long-term effort by the National Cancer Institute and the National Institute of Dental and Craniofacial Research to improve modalities for prevention, early detection, and treatment of oral cancers. This is a natural history study designed to identify markers or early malignant transformation that potentially could be used in predicting which oral soft tissues are most likely to lead to oral cancer.

Persons with white, red, or red/white oral mucosal lesions seen at six Veterans Affairs hospitals in the United States will be selected for the study. Study subjects will undergo a biopsy of all suspect oral lesions. At this baseline examination, the patient will complete a consent form and a questionnaire which will obtain data on potential modifiers of the relationship between histopathology and molecular marker status such as sociodemographic characteristics, tobacco and alcohol use, and medical history. A clinician will describe and photograph the lesion. In addition, the mucosa will be gently scraped to obtain buccal cells. Selected data on dental and medical characteristics of study subjects will be extracted from computerized VA hospital data bases. Biopsy specimens will be analyzed using immunohistochemical and molecular biological approaches to describe their pathological status and to assess the presence of specific molecular events. The analysis of molecular markers may include tests of the presence or activity of certain molecules thought to be associated with the malignant phenotype including p53-dependent growth suppressors, pRb-dependent growth control factors, growth factor receptor-modulated pathways, carcinogen-metabolizing alleles and functioning, and viral agents. To ensure that the best possible scientific paradigm for early malignant changes is tested using this study population, decisions about which genetic and immunohistological assays to conduct on the biopsy material will be made by consensus of the principal and coinvestigators at the time that an adequate sample size is achieved. When biological assays are complete, statistical analysis will determine associations between molecular markers from the oral lesions and the lesions' histopathology and will examine how environmental, behavioral, and sociodemographic factors influence these associations.

Study subjects will then be followed longitudinally over a two-year period to ascertain recurrence of lesions. These study subjects will be asked to return to the dental clinics every 4 months during the first year of the study and every 6 months during the second year. At each visit the patient will receive the same oral examination as at baseline. The patient will be classified as having normal-appearing mucosa or an oral lesion. If a lesion is present, it will be evaluated and characterized as at the baseline and then biopsied. Patients not returning on schedule will be traced, contacted and asked to return for an evaluation. Changes in histopathology and the relationship of these changes to changes in biomarker levels will be examined.

Subjects will be informed that if a gene or genetic change that might be useful for patients with oral lesions is identified, they will be contacted to see whether they would like to have information on which gene types may be associated with oral cancer risk. At that time, prior to making a decision, they will be informed of the various risks and consequences of obtaining such information.

After 14 years, development of new lesions will be identified through 2020 through medical and 3 dental record review and patients vital status and cause of death will be ascertained.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients with white, red, or white and red lesions in the oral cavity and oropharynx as identified by the participating dentist.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons seen at dental clinics at 6 Veterans Affairs Medical Centers who had clinically visible oral lesions@@@
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 1996-08-28 (Actual); Primary Completion 2006-10-04 (Actual); Study Completion 2025-07-29 (Actual)

PRIMARY OUTCOMES:
New or re-emergence of oral lesion | Annually
  the natural history of the oral lesions was assessed via clinical examination over a period of 4 years
oral cancer diagnosis | Once
  Assessed via medical record

CONTACTS AND LOCATIONS:
Overall Officials: Eva Szabo, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (6):
- United States (6):
  - U.C.S.F./ Vterans Affairs Medical Center, San Francisco, California
  - VA Medical Center, Washington D.C., Washington D.C., District of Columbia
  - VA Medical Ctr, Atlanta, Atlanta, Georgia
  - Veterans Affairs, Danville, Danville, Illinois
  - VA Medical Center, Durham, Durham, North Carolina
  - Veterans Affairs, San Antonio, San Antonio, Texas

REFERENCES:
- [Background] Bouquot JE, Gorlin RJ. Leukoplakia, lichen planus, and other oral keratoses in 23,616 white Americans over the age of 35 years. Oral Surg Oral Med Oral Pathol. 1986 Apr;61(4):373-81. doi: 10.1016/0030-4220(86)90422-6. PMID 3458148
- [Background] Brachman DG, Graves D, Vokes E, Beckett M, Haraf D, Montag A, Dunphy E, Mick R, Yandell D, Weichselbaum RR. Occurrence of p53 gene deletions and human papilloma virus infection in human head and neck cancer. Cancer Res. 1992 Sep 1;52(17):4832-6. PMID 1324797
- [Background] Brennan JA, Boyle JO, Koch WM, Goodman SN, Hruban RH, Eby YJ, Couch MJ, Forastiere AA, Sidransky D. Association between cigarette smoking and mutation of the p53 gene in squamous-cell carcinoma of the head and neck. N Engl J Med. 1995 Mar 16;332(11):712-7. doi: 10.1056/NEJM199503163321104. PMID 7854378